CLINICAL TRIAL: NCT00005744
Title: Increased Physical Activity in African-American Women
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4968; R29HL056968 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2004-08

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

SUMMARY:
To conduct a randomized demonstration and education trial of churches in East Baltimore testing a self-help, minimal intervention compared with an intensive physical activity intervention.

DETAILED DESCRIPTION:
BACKGROUND:

The study filled an existing gap by examining how a culturally sensitive physical activity intervention conducted in a community setting was associated with increased daily energy expenditure in African American women -- a group of women who are sedentary and at risk for health problems for which regular physical activity can provide benefits.

DESIGN NARRATIVE:

An evaluation was conducted of the effectiveness of a six-month moderate-intensity physical activity intervention for increasing total daily energy expenditure of sedentary African-American women who were between the ages of 50 and 70 years. The goal of the intervention was to increase total daily energy expenditure by 150 kilocalories per day and time spent in moderate-intensity physical activity by 30 minutes per day. Effects of increased physical activity on selected cardiovascular risk factors (e.g., peak oxygen uptake, blood pressure, HDL cholesterol, serum insulin and plasma glucose) were also determined. Six churches were randomized into intensive or minimal intervention status, and 33 women per church were recruited, for a total of 100 women in each condition. The physical activity intervention consisted of twice-weekly aerobics classes conducted at the churches and additional group-and home-based programming. Volunteer lay leaders were trained as neighborhood exercise specialists to supplement certified aerobics instructors in conducting the intervention.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1996-09; Study Completion 2001-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Young — Johns Hopkins University

REFERENCES:
- [Background] Young DR, Gittelsohn J, Charleston J, Felix-Aaron K, Appel LJ. Motivations for exercise and weight loss among African-American women: focus group results and their contribution towards program development. Ethn Health. 2001 Aug-Nov;6(3-4):227-45. doi: 10.1080/13557850120078143. PMID 11696933
- [Background] Young DR, Jee SH, Appel LJ. A comparison of the Yale Physical Activity Survey with other physical activity measures. Med Sci Sports Exerc. 2001 Jun;33(6):955-61. doi: 10.1097/00005768-200106000-00015. PMID 11404661
- [Background] Young DR, King AC, Sheehan M, Stefanick ML. Stage of motivational readiness: predictive ability for exercise behavior. Am J Health Behav. 2002 Sep-Oct;26(5):331-41. doi: 10.5993/ajhb.26.5.2. PMID 12206443